CLINICAL TRIAL: NCT01546961
Title: The Population Pharmacokinetics of Chloroquine for the Treatment of Uncomplicated P.Vivax Malaria in Pre- and Post-partum Women.
Brief Title: Chloroquine Population Pharmacokinetics in Pre and Post-partum Women
Acronym: KCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMRU1003
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Vivax Malaria
Keywords: Chloroquine; Uncomplicated vivax malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chloroquine (Experimental): Chloroquine phosphate GPO® (Government Pharmaceutical Organization, Thailand) 250 mg (equivalent to chloroquine base 150 mg).
  Dosing will be at 0, 24, 48 hrs with 10 mg/kg on day 0 and day 1, and 5 mg/kg on day 2.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — Chloroquine phosphate GPO® (Government Pharmaceutical Organization, Thailand) 250 mg (equivalent to chloroquine base 150 mg).
  Dosing will be at 0, 24, 48 hrs with 10 mg/kg on day 0 and day 1, and 5 mg/kg on day 2.

SUMMARY:
For the treatment of P.vivax the standard treatment is chloroquine. There is a growing body of evidence suggesting that pregnant women may require different doses of drugs, including antimalarials due to the physiological changes of pregnancy. It is important that any drug used in pregnant women it is given at the correct dose. The only way to evaluate this is by pharmacokinetic studies. The investigators propose to evaluate the pharmacokinetics of chloroquine when use to treat P.vivax in the 2nd or 3rd trimester of pregnancy. The same evaluation in the same woman post-partum is required as a control.

DETAILED DESCRIPTION:
For the treatment of P.vivax the standard treatment is chloroquine. There is a growing body of evidence suggesting that pregnant women may require different doses of drugs, including antimalarials, due to the physiological changes of pregnancy. It is important that any drug used in pregnant women is given at the correct dose. The only way to evaluate this is by pharmacokinetic studies. We propose to evaluate the pharmacokinetics of chloroquine when use to treat P.vivax in the 2nd or 3rd trimester of pregnancy. The same evaluation in the same woman post-partum is required as a control.

The two most recent pharmacokinetic publications conclude differently on chloroquine dosing in pregnant women: one suggests no dose adjustment and the other that a higher dose is probably needed. It is crucial that pregnant women are dosed correctly to maximise cure and minimize the chance for recurrence and the harmful effects of malaria. The proposed study on the pharmacokinetics of chloroquine treatment in pregnant women will solve this dilemma.

Pregnant women on the Thai-Burmese border are encouraged to attend antenatal care often for early detection and treatment of malaria. Low birth weight due to P.vivax affects primigravida and multigravida, not just primarily primigravida as with P.falciparum(highlighted in the attached reference). Hence it is important to consider these women for radical cure. This is not possible during pregnancy as primaquine is contraindicated so the next best time is in the post-partum period. During the post-partum period the woman remains in close contact with midwives for infant care and for their personal health. The midwives also have a record of malaria attacks during pregnancy.

We know more about chloroquine than any other antimalarial used in pregnancy. It has been widely used for prevention and treatment of malaria in pregnancy and in women with autoimmune disease such systemic lupus and rheumatoid arthritis high doses of hydroxychloroquine have been given daily including during the first trimester of pregnancy. Although data from prospective clinical trials of malaria are limited, this drug is considered safe in all trimester of pregnancy and in lactation.

For treatment of uncomplicated P.vivax WHO recommends chloroquine and primaquine where P.vivax remains chloroquine sensitive. A 14 day course of primaquine is recommended for radical cure of P.vivax. WHO advises not to use primaquine during pregnancy or in severe G6PD. WHO permits the use of primaquine during lactation if the breast fed infant is not G6PD deficient.

The possibility that women with recurrent P.vivax in the same pregnancy may have chloroquine resistant P.vivax needs to be considered. While the combination of chloroquine and primaquine cannot be used in pregnancy and the safety and efficacy of ACTs are still undergoing evaluation we need to explore alternatives to chloroquine for such cases. ACTs are recommended for chloroquine resistant P.vivax by WHO and one ACT considered safe in pregnancy and lactation is a 7 day course of artesunate-clindamycin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Gestational age (ultrasound confirmed) > 13.0 weeks
* Viable fetus as assessed by ultrasound scanning
* Microscopically confirmed uncomplicated P.vivax malaria
* Willingness and ability to comply with the study protocol for the duration of the trial
* Written informed consent provided
* No signs of labour

Exclusion Criteria:

* Known hypersensitivity to chloroquine
* Clinical or laboratory features of severe malaria based on WHO criteria-Appendix 1
* Gastrointestinal dysfunction that could alter absorption or motility
* History or known liver diseases or other chronic diseases (excluding thalassaemia & G6PD deficiency)
* Presence of intercurrent illness or any condition which in the judgement of the investigator would place the patient at undue risk or interfere with the results of the study
* Splenectomy
* Hematocrit (HCT) < 20% (based on field reading i.e. capillary sample)
* Taking contraindicated medications
* History of narcotic or alcohol abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Population Pharmacokinetics of Chloroquine | 63 days
  Population pharmacokinetic parameters up to day 63 in pregnant women with uncomplicated P.vivax malaria, and in the same women post-partum with P.vivax or without P.vivax.

SECONDARY OUTCOMES:
Relationship between pharmacokinetics and symptoms | 63 days
  Chloroquine pharmacokinetics versus symptomatology
Efficacy of Chloroquine | 63 days
  Chloroquine efficacy against P.vivax
Reticulocyte counts | 63 days
  Effect of chloroquine treatment on reticulocyte counts
Pregnancy outcomes | 63 days
  Pregnancy outcomes (abortions, low birth weight, premature birth, congenital abnormality, stillbirths, neonatal and infant mortality)

CONTACTS AND LOCATIONS:
Overall Officials: Rose McGready, MD, Principal Investigator — University of Oxford
Locations (1):
- Shoklo Malaria Research Unit, Tak, Mae Sot, Thailand